CLINICAL TRIAL: NCT04997395
Title: Safety and Tolerability of Full Spectrum Cannabidiol Dominant Medicinal Cannabis in Treating Symptoms Associated With Long COVID: A Feasibility Study
Brief Title: Feasibility of Cannabidiol for the Treatment of Long COVID
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bod Australia (Industry)
Collaborators: Drug Science, UK (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BOD202102U; 2021-004534-11 (EudraCT Number)
Record Dates: First submitted 2021-07-31; First posted 2021-08-09 (Actual); Last update posted 2023-01-19 (Actual); Status verified 2023-01

CONDITIONS: Long COVID
Keywords: long COVID; COVID; cannabidiol; post-COVID-19 syndrome; post-COVID syndrome
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- MediCabilis Cannabis sativa 50 (Experimental): The medicinal cannabis used for this study is MediCabilis Cannabis sativa 50, a full spectrum CBD dominant plant based medicinal cannabis containing 50 mg/ml CBD and 2 mg/ml THC.
  On commencing the oral medication, it will be titrated over a 2 week period to a dose of 1 ml twice a day (total dose 2 ml = 100 mg CBD and 4 mg THC). Participants will be given a written titration schedule at the initial clinic visit. There will be the potential for a further dose increase to a total dose of 3 ml per day (150 mg CBD and 6 mg THC) at the 1-month follow-up visit.
  Interventions: Drug: MediCabilis Cannabis sativa 50

INTERVENTIONS:
Drug: MediCabilis Cannabis sativa 50 — Already described
  Other Names: MediCabilis 5%

SUMMARY:
This is an open label, phase 2 clinical trial to assess the feasibility of a cannabidiol (CBD) dominant medicinal cannabis for the treatment of Long COVID. The primary aim is to assess the feasibility of recruiting and retaining individuals diagnosed with Long COVID into a treatment trial of medicinal cannabis, as well as assessing the safety and tolerability of a dominant medicinal cannabis in this population. The secondary aim is to determine the effect of a CBD dominant medicinal cannabis on symptoms associated with Long COVID.

DETAILED DESCRIPTION:
Long COVID, also defined as post-COVID-19 syndrome, is a common outcome after infection with the SARS-COV-2 virus. The need for treatment and ongoing support for people experiencing Long COVID has been increasingly recognised, including through the establishment of dedicated treatment units within the NHS. While symptoms and their severity may vary greatly between individuals, some of the common symptoms associated with Long COVID include fatigue, breathlessness, pain, sleep disturbances and dysautonomia. In this study, we will test the feasibility of a broad spectrum cannabidiol (CBD) dominant formulation, MediCabilis Cannabis sativa 50, for treating these symptoms in people with a diagnosis of Long COVID. CBD is the primary non-psychoactive ingredient in cannabis, and it is being increasingly used in the treatment of symptoms which are similar to those associated with Long COVID. Additionally, there is some evidence that CBD may be effective in reducing inflammation associated with COVID infection. Together, this evidence suggests that it is possible that CBD may be an effective treatment for people diagnosed with Long COVID. We will therefore conduct a feasibility trial in which 30 people are prescribed CBD dominant medical cannabis. Patients will take this medication daily for a total of 21 weeks (2-week titration period, 18-weeks steady dose, 1-week dose reduction), followed by 3-weeks with no medication. We will collect monthly self-report assessments of common symptoms including breathlessness, fatigue, mood, cognition and pain via a smartphone app, as well as real-time data on heart rate, physical activity and sleep using wearable technology. We will also collect daily self-report assessments of key symptoms (mood, pain, fatigue and breathlessness) via a smartphone app for 7 days per 28 days. Our study will establish whether it is feasible to recruit and retain patients with a diagnosis of Long COVID into a trial of a CBD dominant medical cannabis. We will also monitor whether there are any side effects to assess the safety and tolerability of a CBD dominant medical cannabis. Our results will determine the feasibility of medicinal cannabis in the treatment of Long COVID and whether it is safe to use.

ELIGIBILITY:
Inclusion Criteria:

1. Male and females aged 18 years old or above.
2. Long COVID diagnosis, confirmed by either GP triage clinic or attendance and assessment by a Long COVID clinic. Self-diagnosed Long COVID will not be included in the study. It is expected that in order to have a coded diagnosis of long Covid, the participant will have undertaken the relevant clinical assessment and investigations as recommended by the NICE guidance on Long COVID. https://www.nice.org.uk/guidance/ng188
3. Females must be non-pregnant, non-lactating.
4. Proficient in English and have internet access and a mobile phone.
5. Stated willingness to comply with all study procedures and availability for the duration of the study.
6. Provision of signed and dated informed consent form.
7. All male and females of childbearing potential must agree to use highly effective contraception from the time of signing informed consent until 3 months (12 weeks) after the treatment has stopped. Participants using systemically acting hormonal contraception for example the oral contraceptive pill or contraceptive implant should use an additional non-hormonal/reliable barrier method of contraception from the time of signing informed consent until 3 months (12 weeks) after the treatment has stopped.

Exclusion Criteria:

1. Self-diagnosed Long COVID without relevant assessment and investigation as per clinical guidelines.
2. Serious ongoing medical and/or psychiatric illnesses/disorders that will require active and variable treatment during the trial period. (this will be assessed from clinical history and GP records)
3. Used cannabinoids or a cannabinoid-based medicine within 3 months prior to study Day 1 and unwillingness to abstain from recreational drug use during the study period.
4. Cannabis dependence or any other drug or alcohol dependence within the past two years.
5. Known hypersensitivity to cannabis-based products or any of the excipients in the study drug.
6. Use of any other investigational products within 30 days of screening day.
7. Use of anti-coagulant drugs such as warfarin.
8. History of attempted suicide, bipolar disorder or schizophrenia.
9. History of chronic liver failure or present history of an abnormal liver function (LFT) blood test within the 3 months prior to recruitment. This should be able to be confirmed during the screening process as all participants should have had a liver function blood test as part of the recommended clinical assessment prior to diagnosing Long COVID. If no liver function test is available within 6 months of screening (which is unlikely), participants will be asked if they would agree to having a screening LFT.
10. History of allergy to tree nuts, with no definite previous coconut exposure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2022-04-14 (Actual); Primary Completion 2023-01-06 (Actual); Study Completion 2023-01-06 (Actual)

PRIMARY OUTCOMES:
Recruitment rate | 12 months (48 weeks)
  Recruiting individuals diagnosed with long COVID into a treatment trial of medicinal cannabis
Tolerability for the treatment of long COVID | 6 months (24 weeks)
  Retaining participants in a six month trial of medicinal cannabis using the proposed battery of assessments. Retention rate (%) of participants enrolled into the trial who complete the six-month protocol.
Number of side effects | 6 months (24 weeks)
  Adverse events, side effects

SECONDARY OUTCOMES:
Long COVID symptoms | 5 months (20 weeks)
  Assessed by the COVID-19 Yorkshire Rehabilitation Scale (C19-YRS, Sivan et al., 2021). This scale includes: breathlessness, cough/ voice, swallowing/ nutrition, fatigue, continence, cognition, pain/discomfort, anxiety, depression, post-traumatic stress disorder, communication, mobility, personal care, activities of daily living, social role, perceived health status and family/carers views. The C19-YRS provides an overview of 3 outcomes: symptoms severity score, functional disability score and global health score.
Fatigue | 5 months (20 weeks)
  Fatigue will be assessed using the nine item Fatigue Severity Scale (Krupp et al., 1989). This scale, which was initially designed for use in multiple sclerosis and systemic lupus erythematosus has been used extensively across multiple disorders and has bene demonstrated to have good reliability and validity. Each of the nine items in this scale is assessed on a seven-point scale from 1 (strongly disagree) to 7 (strongly agree). Thus, the composite scale ranges from 9 to 63 with higher ratings representing more severe fatigue.
Self-reported quality of life | 5 months (20 weeks)
  The health-related quality of life instrument that will be used in this study is the EuroQol 5 Dimensions (EQ-5D; Devlin et al., 2017). It is a widely used, validated, and reliable tool that assesses the quality of life of patients in many disease areas through assessment of the severity of each of 5 dimensions (mobility, self-care, usual activities, pain/discomfort and anxiety/depression). Each dimension has 5 levels (1-5): no problems, slight problems, moderate problems, severe problems and extreme problems. The digits for the five dimensions can be numerically summed into a single number, varying from 5 to 25 with higher numbers representing a lower quality of life. In addition, this measure contains a 100-point visual analogue which asks respondents to rate their current health with higher numbers representing better health.
Pain score | 5 months (20 weeks)
  The Brief Pain Inventory Short Form (BPI-SF; Cleeland, 1989; Cleeland & Ryan, 1994), a 9 item self-administered questionnaire, will be used to evaluate the severity of a patient's pain and the interference of this pain on the patient's daily feeling and functioning. The patient rates their worst, least, average, and current pain intensity, list current treatments and their perceived effectiveness, and rate the degree that pain interferes with general activity, mood, walking ability, normal work, relations with other persons, sleep, and enjoyment of life on a 10-point scale. The BPI scale defines pain as follows: 1-4=Mild Pain, 5-6=Moderate Pain, 7-10=Severe Pain. Thus, a mean of the items can be presented with higher ratings representing more severe pain. In addition, the mean of the 7 items assessing interference, each rated on a scale from 0 to 10, will be used as a measure of mean pain interference with higher numbers representing more interference.
Mood (anxiety) | 5 months (20 weeks)
  The Generalised Anxiety Disorder Assessment (GAD-7; Spitzer et al., 2006) will be used to measure depression. The GAD-7 is a seven-item instrument that is used to measure or assess the severity of generalised anxiety disorder (GAD). Each item asks the individual to rate the severity of their symptoms over the past two weeks. Response options include "not at all", "several days", "more than half the days" and "nearly every day". The GAD-7 score is calculated by assigning scores of 0, 1, 2, and 3, to the response categories of "not at all," "several days," "more than half the days," and "nearly every day," respectively, and then adding together the scores for the seven questions. GAD-7 total score for the seven items ranges from 0 to 21.
Mood (depression) | 5 months (20 weeks)
  The Patient Health Questionnaire (PHQ-9; Kroneke et al., 2001) will be used to measure mood/ depression. It is a reliable and valid measure of depression severity and is comprised of a 9-item self-rated instrument that has been validated in general populations, medical populations and psychiatric samples.
  It is calculated by assigning scores of 0, 1, 2, and 3, to the response categories of not at all, several days, more than half the days, and nearly every day, respectively. PHQ-9 total score for the nine items ranges from 0 to 27.
Sleep quality | 5 months (20 weeks)
  Assessed using Pittsburgh self-report questionnaires and wearable technology. The Pittsburgh Sleep Quality Index (PSQI) includes a scoring key for calculating a patient's seven subscores, each of which can range from 0 to 3. The subscores are tallied, yielding a "global" score that can range from 0 to 21. A global score of 5 or more indicates poor sleep quality; the higher the score, the worse the quality. Mean ratings on this global score will be used in our analyses. Furthermore, the wearable technology (i.e. Fitbit) will provide the patients' total time in sleep and time in sleep stages (light, deep and REM sleep), as well as a daily Sleep Score accessed via the Fitbit app. Seven day averages (means) of the Fitbit measures will be calculated for each participant across the duration of the study.
Resting heart rate (expressed as average beats per minute) | 5 months (20 weeks)
  The wearable technology will provide 24/7 heart rate tracking and heart rate variability. We will have access to the daily resting heart rate and averages across discrete periods. We will analyse mean resting heart rate (beats per minute). Variation in the time between each heartbeat (heart rate variability) will be accessed via the Fitbit app. Seven day averages (means) of the Fitbit measures will be calculated for each participant across the duration of the study.
Activity levels (number of daily steps, distance walked, stairs climbed, active minutes and calories burned) | 5 months (20 weeks)
  Activity levels assessed via wearable technology. The wearable technology (i.e. Fitbit) tracks all-day activity including number of steps walked, distance walked (expressed in kilometres), floors climbed, active minutes and calories burned. We will analyse the seven-day mean number of daily steps, distance walked, stairs climbed, active minutes and calories burned. Seven day averages (means) of the Fitbit measures will be calculated for each participant across the duration of the study.
Oxygen saturation (expressed as percentage saturation) | 5 months (20 weeks)
  Oxygen saturation expressed as percentage saturation, with typical numbers being in the region of 95% will also be assessed via the Fitbit. Seven day averages (means) of the Fitbit measures will be calculated for each participant across the duration of the study.
Daily symptoms | 5 months (20 weeks)
  Assessed using daily reports of key symptoms (breathlessness, fatigue, mood and pain) adapted from the COVID-19 Yorkshire Rehabilitation Scale. Each symptom will be scored out of 10 for a period of 7 days per 28 days, to produce an average score for each symptom.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Iveson, Principal Investigator — Steps Neurorehabilitation Unit
Locations (1):
- Drug Science, York, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: From 12 months after completion of data collection.
Access Criteria: Ethical approval obtained from recognised ethics committee/ IRB Subject to oversight and approval by research team. All identifiers to be removed.